CLINICAL TRIAL: NCT02474134
Title: A Phase 1 Double-Blind, Randomised, Two-Treatment Cross-over Study Comparing the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PF530 and Betaferon Administered by Subcutaneous Injection in Healthy Adult Volunteers
Brief Title: Comparison Study of PF530 and Betaferon in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfenex, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PF530-101
Record Dates: First submitted 2015-03-17; First posted 2015-06-17 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF530/Betaferon (Other): Single subcutaneous injection of two interferon beta-1b products (PF530 and Betaferon) 0.25 mg
  Interventions: Drug: Interferon beta-1b (PF530, Betaferon)
- Betaferon/PF530 (Other): Single subcutaneous injection of two interferon beta-1b products (Betaferon and PF530) 0.25 mg
  Interventions: Drug: Interferon beta-1b (PF530, Betaferon)

INTERVENTIONS:
Drug: Interferon beta-1b (PF530, Betaferon) — Single subcutaneous administration
  Other Names: PF530, Betaferon

SUMMARY:
The purpose of this study is to compare the safety, tolerability, and blood levels of two interferon beta-1b products, Betaferon and PF530, in healthy volunteers.

DETAILED DESCRIPTION:
This is a double-blind, randomised, two-treatment cross-over study in healthy adult subjects to compare the safety, tolerability, pharmacokinetics and pharmacodynamics of PF530 and Betaferon. Half of the subjects will be randomised to receive PF530 first and Betaferon second, and the other half will be randomised to receive the drugs in reverse sequence. Each study participant will complete two 7-day study periods (Period 1 and Period 2), separated by a 14-day washout period. In Part I of the study, 12 subjects will be enrolled for an initial assessment. In Part II, up to 36 additional subjects may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential must agree to use two effective methods of birth control, practice complete abstinence, or confirm sterilization of monogamous male partner
* Males must have had a documented vasectomy, practice complete abstinence or use a condom and refrain from sperm.
* Participant is free from clinically significant illness or disease as determined by medical and surgical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory assessments.
* Able to understand and sign the written Informed Consent Form

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, metabolic, psychological, musculoskeletal disease or malignancies unless deemed not clinically significant by the Principal Investigator.
* Previous treatment with any interferon product, including investigational use.
* Participants with a history of malignant disease, including solid tumours and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
* Positive screening test for human immunodeficiency virus (HIV).
* Positive screening test for hepatitis C antibody (HCV Ab) or current hepatitis B infection (defined as positive for hepatitis surface antigen [HBsAg] at Screening). Participants with immunity to hepatitis B (defined as negative HBsAg and positive hepatitis B surface antibody [HBsAb]) are eligible to participate in the study.
* History of epilepsy, seizure disorder or any unexplained black-outs.
* History of hypersensitivity or intolerance to paracetamol or non-steroidal anti-inflammatory drugs (NSAID) that would preclude the use of at least 1 of these during the study.
* History of severe allergic or anaphylactic reactions or a known allergy to any component of the interferon β-1b formulation.
* History of drug or alcohol abuse less than or equal to 12 months prior to Screening.
* History of tobacco use less than or equal to 6 months prior to Screening.
* A positive test for drugs of abuse or alcohol during Screening or prior to dosing.
* Unwilling or unable to abstain from alcohol from 7 days prior to dosing until end-of-study assessments.
* Use of any prescription medication, over-the-counter medication, or herbal supplements/products during Screening or throughout study, unless approved by both the Principal Investigator and the Sponsor.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) and serious adverse event (SAE) incidence | 28 Days

SECONDARY OUTCOMES:
Serum area-under-the-curve (AUC) of PF530 and Betaferon | 72 hours
Serum maximum concentration (Tmax) of PF530 and Betaferon | 72 hours
Serum half-life (t1/2) of PF530 and Betaferon | 72 hours
Serum neopterin | 168 hours
Serum myxovirus resistance protein A | 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, MD, Principal Investigator — CMAX, A Division of IDT Australia, Limited; Hubert C Chen, MD, Study Director — Pfenex, Inc
Locations (1):
- CMAX, Adelaide, South Australia, Australia